CLINICAL TRIAL: NCT05859607
Title: Predictors of Difficult Laparoscopic Cholecystectomy, Scoring Systems and Their Implications on the Outcomes, Sohag Experience.
Brief Title: Predictors of Difficult Laparoscopic Cholecystectomy, Scoring Systems and Their Implications on the Outcomes , Sohag Experience.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Fahmy Mahmoud, resident doctor at General surgery department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-03-14MS
Record Dates: First submitted 2023-04-03; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Chronic Calculous Cholecystitis
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Easy cholecystectomy (Active Comparator): easy procedure with no complications
  Interventions: Procedure: laparoscopic cholecystectomy
- moderate severe cholecystectomy (Active Comparator): moderate severity with prolonged time or complication .
  Interventions: Procedure: laparoscopic cholecystectomy
- difficult cholecystectomy (Active Comparator): very prolonged time , complication or conversion to open cholecystectomy .
  Interventions: Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy — conventional laparoscopic cholecystectomy with calculation of difficulty scorings

SUMMARY:
laparoscopic cholecystectomy nowadays is the most common surgery done by General surgery surgeons , so it is necessary to evaluate the difficulty of each case prior to surgery and from the first look ,to avoid complications and improve outcomes , so scoring systems are needed for better assessment of the overall condition and make good decision .

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic gall stones

Exclusion Criteria:

* lap to open conversion due to equipment failure pregnancy common bile duct stone obstructive jaundice unfit for general anesthesia patients refusing lap cholecystectomy.

Min Age: 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-10-18 (Estimated); Study Completion 2023-10-18 (Estimated)

PRIMARY OUTCOMES:
Validation and applicability of scoring systems | 6 months
  the scoring system should reach high percentage to be applicable and could be used for scoring difficulty.A comparison between preoperative score and intraoperative score, then the success of a scoring system is by the high percentage sensitivity ,preoperative data sheet will be taken from all patients ,then the first look intraoperative will judge the score through multiple items , the cross matching will be done between the two scores. and to measure the results,There are many scoring system for example Randawa preoperative and intraoperative score , Nassar preoperative and intraoperative score ,matching the result of both preoperative and intraoperative will be done to validate each one. Randawa score classified into easy and moderate and severe difficulty based on time lapsed during cholycystectomy ,intraoperative problems and complications Nassar uses the intraoperative shape of gall bladder to classify the difficulty from 1 to 5 grades upon the first look to the gall bladder.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided